CLINICAL TRIAL: NCT00472888
Title: Clinical Factors Associated With Floppy Iris Signs: a Prospective Study From Two Centers
Brief Title: Clinical Factors Associated Floppy Iris
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Other Study IDs: KA 05/244
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Pupil Constriction; Iris Floppiness; Iris Prolapsus From the Wound
Keywords: Alpha-adrenergic blockers; cataract surgery; pseudoexfoliation syndrome; diabetes mellitus; hypertension; pupil
MeSH Terms: conditions — Miosis; Exfoliation Syndrome; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is planned to investigate the incidence of intraoperative floppy iris and its relationship with pseudoexfoliation, diabetes, hypertension as well as systemic alpha-1 adrenergic blocker use.

DETAILED DESCRIPTION:
Our aim is to investigate the incidence of intraoperative floppy iris syndrome (IFIS) signs and evaluate the relationship of IFIS signs as well as complete IFIS with pseudoexfoliation, diabetes, hypertension, and alpha-1 adrenergic blocker (A1AB) use. Five-hundred patients will be included in this prospective study. Preoperatively, pupil diameter before and after dilation, presence of pseudoexfoliation, history of diabetes, hypertension, and use of any A1AB will be recorded. Intraoperative adverse events such as pupillary constriction, iris billowing, and iris prolapse from the wound will be noted. Multinomial regression analysis will be used to evaluate the relationship of IFIS signs with pseudoexfoliation, diabetes, hypertension, and A1AB usage. According to the results we will determine the incidence of IFIS in our patient population and evaluate its relationship with alpha-1 adrenergic blocker use. We will also investigate the relationship of floppy iris problems with pseudoexfoliation, diabetes, high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the diagnosis of cataract who were decided to have phacoemulsification

Exclusion Criteria:

* Previous history of trauma or surgery of the eye, congenital ocular disease including cataract, infection, inflammation, angle closure glaucoma, or medication (topical) that might affect the size and shape of the pupil

Only the first operated eye of each patient was included.

Ages: 28 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-11; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rana Altan-Yaycioglu, MD, Study Chair — Baskent University, Faculty of Medicine, Department of Ophthalmology; Yonca A Akova, MD, Study Director — Baskent University, Faculty of Medicine, Department of Ophthalmology
Locations (1):
- Baskent University, Faculty of Medicine, Department of Ophthalmology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Chang DF, Campbell JR. Intraoperative floppy iris syndrome associated with tamsulosin. J Cataract Refract Surg. 2005 Apr;31(4):664-73. doi: 10.1016/j.jcrs.2005.02.027. PMID 15899440
- [Background] Schwinn DA, Afshari NA. alpha(1)-Adrenergic receptor antagonists and the iris: new mechanistic insights into floppy iris syndrome. Surv Ophthalmol. 2006 Sep-Oct;51(5):501-12. doi: 10.1016/j.survophthal.2006.06.011. PMID 16950249
- [Derived] Altan-Yaycioglu R, Gedik S, Pelit A, Akova YA, Akman A. Clinical factors associated with floppy iris signs: a prospective study from two centers. Ophthalmic Surg Lasers Imaging. 2009 May-Jun;40(3):232-8. doi: 10.3928/15428877-20090430-02. PMID 19485285